CLINICAL TRIAL: NCT03682783
Title: The Development of Artificial Intelligence-assisted Glaucoma Screening Program
Brief Title: Artificial Intelligence-assisted Glaucoma Screening (AIAGS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Haiyan Wang, Attending of Ophthalmology, M.D. Ph.D., Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 81300776
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Glaucoma Eye
Keywords: Artificial Intelligence; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fundus Image: Glaucomatous and Non-glaucomatous fundus images that have been taken from the last 5 years in Shanghai General hospital.
  Interventions: Diagnostic Test: Fundus Image

INTERVENTIONS:
Diagnostic Test: Fundus Image — Fundus image of optic nerve

SUMMARY:
This study will develop an artificial intelligence (AI) program for the screening of glaucoma.

DETAILED DESCRIPTION:
We have realized that the glaucomatous optic neuropathy is irreversible. But if early detection and early intervention can be performed to control the development of the disease, it can greatly reduce the blindness rate of glaucoma, improve the life quality and physiological and mental health of patients, and alleviate the social burden. Therefore, screening and early diagnosis of glaucoma is the focus of glaucoma prevention.

China has a population of 1.3 billion, which greatly increase the difficulty of disease screening. In recent years, the intersection of artificial intelligence (AI) technology and modern medicine has made efficient and rapid disease screening possible.

ELIGIBILITY:
Inclusion Criteria:

* able to complete fundus images

Exclusion Criteria:

* unable to complete fundus images

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Both glaucoma and non-glaucoma patients who can complete fundus image test will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
The specificity of the algorithm for diagnosing glaucoma | from January 2020 to March 2021
  The specificity of the algorithm for diagnosing glaucoma will be calculated ...
The sensitivity of the algorithm for diagnosing glaucoma | from January 2020 to March 2021
  The sensitivity of the algorithm for diagnosing glaucoma will be calculated .

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wang, Ph.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China